CLINICAL TRIAL: NCT01481259
Title: Maintenance Immunotherapy With Autologous Cytokine-induced Killer Cells for Stage IIIb/IV Nonsquamous Non-small Cell Lung Cancer
Brief Title: Maintenance Therapy With Autologous Cytokine-induced Killer Cells for Nonsquamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Guosheng Feng, Professor, People's Hospital of Guangxi Zhuang Autonomous Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIKLC-201004
Record Dates: First submitted 2011-11-16; First posted 2011-11-29 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Nonsquamous non-small cell lung cancer; Maintenance therapy; Immunotherapy; Autologous cytokine-induced killer cell; Pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immunotherapy (Experimental): Subjects receive autologous cytokine-induced killer cell infusion every 21 days
  Interventions: Biological: Autologous cytokine-induced killer cell
- Pemetrexed (Active Comparator): Subjects receive pemetrexed infusion at a dose of 500mg/m2 every 21 days
  Interventions: Other: Pemetrexed

INTERVENTIONS:
Biological: Autologous cytokine-induced killer cell — Subjects receive autologous cytokine-induced killer cell infusion every 21 days in the absence of disease progression or unacceptable toxicity.
  Arms: Immunotherapy
Other: Pemetrexed — Subjects receive pemetrexed infusion at a dose of 500mg/m2 every 21 days in the absence of disease progression or unacceptable toxicity.
  Arms: Pemetrexed

SUMMARY:
Maintenance therapy has been considered as an important component to prolong survival in patients with advanced Nonsquamous Non-small Cell Lung Cancer (NSCLC). Previous studies have confirmed that pemetrexed is one of the effective drugs in improving progression-free survival for stage IIIb-IV nonsquamous non-small cell lung cancer. With the periodic deliveries of pemetrexed, however,the functioning status and immune system may get worse, which subsequently has an negative impact on patient's quality-of-life. Immunotherapy with autologous cytokine-induced killer (CIK) cells can activate the antitumor defense mechanism through stimulating immune response and altering the interaction between tumor and its host. This effect may result in improved tumor control and survival, as well as a better quality of life. To test the hypothesis, a randomised controlled study was conducted to compare CIK cells with pemetrexed as maintenance therapy for stage IIIb-IV nonsquamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven nonsquamous non-small cell lung cancer
* Stage IIIb-IV, according to AJCC 2010 Staging System
* Disease measurable
* Patients are currently receiving two-drug chemotherapy regimen containing a platinum-based drug as first-line therapy
* No chemotherapy or radiotherapy prior to first-line therapy
* Age between 18-75
* Performance status <2
* No congestive heart failure, severe arrhythmia,and coronal atherosclerosis heart disease
* No uncontrolled metabolic disease, infection, and neurological disorders
* No other malignancies
* Signed study-specific consent form prior to study entry

Exclusion Criteria:

* Patients are currently receiving radiotherapy or any chemotherapy regimen other than two-drug containing a platinum-based drug as first-line therapy
* Pregnant or lactating women
* Patient having hepatitis B virus infection, active tuberculosis, or other infectious diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | One year

SECONDARY OUTCOMES:
Overall survival | Two years
Toxicities | Two years
Quality-of-life | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Guosheng Feng, M.D, Principal Investigator — People's Hospital of Guangxi Zhuang Autonomous Region; Hui Lin, M.D, Study Chair — People's Hospital of Guangxi Zhuang Autonomous Region; Yuan Liang, M.D, Study Chair — Guangxi Department of Public Health; Heming Lu, M.D, Study Chair — People's Hospital of Guangxi Zhuang Autonomous Region
Locations (1):
- Clinical Cancer Center, People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi, China